CLINICAL TRIAL: NCT02248571
Title: An Open Label, randomIzed Controlled Prospective Multicenter Two Arm Phase IV Trial to Determine Patient Preference for Everolimus in Combination With Exemestane or Capecitabine in Combination With Bevacizumab for Advanced (Inoperable or Metastatic) HER2-negative Hormone Receptor Positive Breast Cancer
Brief Title: Patient Preference for Everolimus in Combination With Exemestane or Capecitabine in Combination With Bevacizumab
Acronym: IMPROVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: iOMEDICO AG (Industry)
Collaborators: Arbeitsgemeinschaft fur Internistische Onkologie (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: iOM-12293
Record Dates: First submitted 2014-08-28; First posted 2014-09-25 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer Recurrent; HER2/Neu-negative Carcinoma of Breast; Hormone Receptor Positive Malignant Neoplasm of Breast
Keywords: breast cancer; advanced; inoperable; metastatic; HER2/neu-negative; hormone receptor positive; HR+; female; postmenopausal
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Bevacizumab; Capecitabine; Everolimus; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Bevacizumab plus Capecitabine (1st treatment phase) followed by Everolimus plus Exemestane (2nd treatment phase)
  Dosing (treatment cycle: 21days):
  1. Capecitabine: 1000 mg/m2 orally applied twice daily as combined 150 mg and 500 mg tablets on days 1 to 14 of each 21-day cycle, followed by a seven day rest period (i.e. off-treatment) --- Bevacizumab: 15 mg/kg intravenously applied once every three weeks (i.e. 5 mg/kg/wk dose equivalent)
  2. Everolimus: 10 mg/day orally applied tablet --- Exemestane: 25 mg/day orally applied tablet
  Patient questionaires to assess patient reported outcome and patients' preference will be completed at four specific time points during study treatment (two timepoints in each treatment phase)
  Interventions: Drug: Bevacizumab; Drug: Capecitabine; Drug: Everolimus; Drug: Exemestane; Other: Patient questionaires
- Arm B (Experimental): Everolimus plus Exemestane (1st treatment phase) followed by Bevacizumab plus Capecitabine (2nd treatment phase)
  Dosing (treatment cycle: 21days):
  1. Everolimus: 10 mg/day orally applied tablet --- Exemestane: 25 mg/day orally applied tablet
  2. Capecitabine: 1000 mg/m2 orally applied twice daily as combined 150 mg and 500 mg tablets on days 1 to 14 of each 21-day cycle, followed by a seven day rest period (i.e. off-treatment) --- Bevacizumab: 15 mg/kg intravenously applied once every three weeks (i.e. 5 mg/kg/wk dose equivalent)
  Patient questionaires to assess patient reported outcome and patients' preference will be completed at four specific time points during study treatment (two timepoints in each treatment phase)
  Interventions: Drug: Bevacizumab; Drug: Capecitabine; Drug: Everolimus; Drug: Exemestane; Other: Patient questionaires

INTERVENTIONS:
Drug: Bevacizumab — administered as combined therapy with Capecitabine
  Other Names: Avastin®
Drug: Capecitabine — administered as combined therapy with Bevacizumab
Drug: Everolimus — administered as combined therapy with Exemestane
  Other Names: Afinitor®
Drug: Exemestane — administered as combined therapy with Everolimus
Other: Patient questionaires — Patients will fill out questionaires at four specific time points during study treatment to assess patient reported outcome and patients' preference
  Other Names: Papient reported outcome; Patients' preference

SUMMARY:
This is a clinical trial with a crossover design to determine patients' preference for capecitabine in combination with bevacizumab or everolimus in combination with exemestane for advanced breast cancer patients and to evaluate, if any combination is associated with a better quality of life.

To identify patients' preference for either therapy in this trial, patients without disease progression or other reasons for early discontinuation will be asked for their treatment preference and their treatment satisfaction. To correlate patients' preference with other patient reported outcomes (PROs), quality of life (QoL) will be assessed at baseline and throughout the study, using dedicated questionnaires.

With similarly active treatment options, it is of utmost importance to identify the treatment that has the least negative impact on the patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent must be obtained prior to any study specific procedure.

1. Adult women (≥ 18 years of age)
2. . Postmenopausal status

   The investigator must confirm postmenopausal status. Postmenopausal status is defined either by:
   * Age ≥ 55 years and one year or more of amenorrhea
   * Age < 55 years and one year or more of amenorrhea and postmenopausal levels of follicle stimulating hormone (FSH) and Luteinizing hormone (LH) per local institutional standards
   * Prior hysterectomy and has postmenopausal levels of FSH and LH per local institutional standards
   * Surgical menopause with bilateral oophorectomy
   * For women with therapy-induced amenorrhea, oophorectomy or serial measurements of FSH and / or estradiol are needed to ensure postmenopausal status.

   Note: Ovarian radiation or treatment with a luteinizing hormone-releasing hormone (LH-RH) agonist (goserelin acetate or leuprolide acetate) is not permitted for induction of ovarian suppression.
3. Pathologically confirmed HER2/neu-negative, ER/PR positive inoperable or metastatic adenocarcinoma of the breast
4. Indication for systemic palliative targeted therapy / first line chemotherapy after failure of at least one non-steroidal aromatase inhibitor therapy at any time during the disease course (no restriction regarding the number of previous endocrine lines)
5. No indication for other chemotherapeutic treatment including Taxanes or Anthracyclines
6. Measurable or non-measurable disease as per RECIST 1.1
7. Adequate bone marrow, liver and renal function (according to current SmPCs of both treatment regimens)
8. ECOG performance status 0-2
9. Fluent German (spoken and written) language

Exclusion Criteria:

1. Prior palliative cytotoxic chemotherapies
2. Prior exposure to mTOR-Inhibitors (prior treatment with exemestane is allowed)
3. Concomitant antihormonal therapies, other than study medication
4. Symptomatic visceral metastases (as deemed by the investigator)
5. Uncontrolled CNS metastases
6. Unstable skeletal metastases
7. Medically uncontrolled cardiovascular diseases (e.g. uncontrolled hypertension)
8. Medically uncontrolled diabetes mellitus
9. Severe hepatic impairment (Child-Pugh C)
10. Inadequate organ function as specified below:

    * Hemoglobin < 9.0 g/dl
    * Absolute neutrophil count (ANC) <1,5 x109/L
    * Platelets <100 x109/L
    * Creatinine clearance < 30ml/min [Cockcroft and Gault]
11. Known HIV infection or chronic hepatitis B or C or history of hepatitis B or C
12. Known dihydropyrimidine dehydrogenase (DPD) deficiency
13. Any other contraindications to the study drugs used or their excipients according to current SmPCs
14. Concomitant use of immunosuppressive agents or chronic use of systemic corticosteroids
15. Use of any other concomitant medication known to interfere with the study drugs
16. Use of concomitant medication known to interfere with the study results (e.g. hormonal therapy) during the whole study duration
17. Premenopausal patients
18. Pregnant or breast feeding patients
19. Participation in additional parallel interventional drug or device studies within four weeks before start of study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Patients' preference | After 12 weeks of second treatment phase or two weeks after early (< 12 weeks) treatment discontinuation
  Patients' preference of the two treatment combinations capecitabine plus bevacizumab or everolimus in combination with exemestane after failure of standard antihormonal therapy in patients with advanced (inoperable or metastatic) HER2/neu-negative hormone receptor positive breast cancer.
  The preference will be ascertained using the patient preference questionnaire.

SECONDARY OUTCOMES:
Reasons for patients' preference | After 12 weeks of second treatment phase or two weeks after early (< 12 weeks) treatment discontinuation
  To evaluate reasons for preference as assessed by the patient preference questionnaire
Patient reported treatment satisfaction | After 12 weeks of first and second treatment phase or two weeks after early (< 12 weeks) treatment discontinuation of each treatment phase
  To compare patient reported treatment satisfaction as assessed by the treatment satisfaction questionnaire in first- and second treatment phase
Quality of life | At baseline and after 12 weeks of first and second treatment phase or two weeks after early (< 12 weeks) treatment discontinuation of each treatment phase
  To investigate differences in quality of life by the European Organization for Research and Treatment of Cancer quality of life questionnaire 30 (EORTC QLQ-C30) and EORTC QLQ-FA13 questionnaire
Progression free survival rate | After 12 weeks of first and second treatment phase
  To assess progression free survival rates after 12 weeks of therapy in first- (PFS rate 1) and second treatment phase (PFS rate 2)
Objective response rates and disease control rates based on tumor assessment (RECIST 1.1) | Participants will be followed for the whole duration of first phase therapy, with an expected average of 12 months, plus 3 months of second phase therapy (15 months in total)
  To assess clinical benefit by determining objective response rates and disease control rates based on tumor assessment as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
Safety and tolerability as measured by number of treatment-emergent adverse events (AEs) and clinical laboratory abnormalities | From date of informed consent to +30 days from last application of study medication
  To evaluate safety and tolerability throughout the study according to Common Toxicity Criteria for Adverse Effects (CTCAE) 4.03 criteria, including clinical laboratory (grades 3 or 4 - separately for hematology and biochemistry) and number of treatment-emergent AEs (safety data for pre- and post-treatment periods will be listed separately)
Physicians' treatment preference | After 12 weeks of second treatment phase or two weeks after early (< 12 weeks) treatment discontinuation
  To determine physicians' treatment preference as assessed by the physician preference questionnaire
Progression free survival for first and second treatment phase | Participants will be followed until progressive disease in boths treatment phases (expected 21 months in total)
  To explore progression free survival separately for each treatment phase
Overall survival | Participants will be followed until death (expected median of 24 months)
  To explore overall survival for each treatment arm beginning from start of respective treatment phase until end of follow-up phase

OTHER OUTCOMES:
Relationship Quality of life scores / patient preference | At baseline and after 12 weeks of first and second treatment phase or two weeks after early (< 12 weeks) treatment discontinuation of each treatment phase
  To explore relationship between QoL scores and patient preference (Exploratory objective)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Decker, MD, Principal Investigator — practice based oncology office Ravensburg
Locations (1):
- iOMEDICO AG, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baselga J, Campone M, Piccart M, Burris HA 3rd, Rugo HS, Sahmoud T, Noguchi S, Gnant M, Pritchard KI, Lebrun F, Beck JT, Ito Y, Yardley D, Deleu I, Perez A, Bachelot T, Vittori L, Xu Z, Mukhopadhyay P, Lebwohl D, Hortobagyi GN. Everolimus in postmenopausal hormone-receptor-positive advanced breast cancer. N Engl J Med. 2012 Feb 9;366(6):520-9. doi: 10.1056/NEJMoa1109653. Epub 2011 Dec 7. PMID 22149876
- [Background] Yardley DA, Noguchi S, Pritchard KI, Burris HA 3rd, Baselga J, Gnant M, Hortobagyi GN, Campone M, Pistilli B, Piccart M, Melichar B, Petrakova K, Arena FP, Erdkamp F, Harb WA, Feng W, Cahana A, Taran T, Lebwohl D, Rugo HS. Everolimus plus exemestane in postmenopausal patients with HR(+) breast cancer: BOLERO-2 final progression-free survival analysis. Adv Ther. 2013 Oct;30(10):870-84. doi: 10.1007/s12325-013-0060-1. Epub 2013 Oct 25. PMID 24158787
- [Background] Miller KD, Chap LI, Holmes FA, Cobleigh MA, Marcom PK, Fehrenbacher L, Dickler M, Overmoyer BA, Reimann JD, Sing AP, Langmuir V, Rugo HS. Randomized phase III trial of capecitabine compared with bevacizumab plus capecitabine in patients with previously treated metastatic breast cancer. J Clin Oncol. 2005 Feb 1;23(4):792-9. doi: 10.1200/JCO.2005.05.098. PMID 15681523
- [Background] Robert NJ, Dieras V, Glaspy J, Brufsky AM, Bondarenko I, Lipatov ON, Perez EA, Yardley DA, Chan SY, Zhou X, Phan SC, O'Shaughnessy J. RIBBON-1: randomized, double-blind, placebo-controlled, phase III trial of chemotherapy with or without bevacizumab for first-line treatment of human epidermal growth factor receptor 2-negative, locally recurrent or metastatic breast cancer. J Clin Oncol. 2011 Apr 1;29(10):1252-60. doi: 10.1200/JCO.2010.28.0982. Epub 2011 Mar 7. PMID 21383283
- [Background] Escudier B, Porta C, Bono P, Powles T, Eisen T, Sternberg CN, Gschwend JE, De Giorgi U, Parikh O, Hawkins R, Sevin E, Negrier S, Khan S, Diaz J, Redhu S, Mehmud F, Cella D. Randomized, controlled, double-blind, cross-over trial assessing treatment preference for pazopanib versus sunitinib in patients with metastatic renal cell carcinoma: PISCES Study. J Clin Oncol. 2014 May 10;32(14):1412-8. doi: 10.1200/JCO.2013.50.8267. Epub 2014 Mar 31. PMID 24687826